CLINICAL TRIAL: NCT06587958
Title: Fermented Plant-based Portfolio Diet 4 Metabolic Health (FermDiHealth)
Brief Title: Fermented Plant-based Portfolio Diet 4 Metabolic Health
Acronym: FermDiHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chalmers University of Technology (Other)
Collaborators: KU Leuven (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Rikard Landberg, Professor, Chalmers University of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Chalmers-FermDiHealth
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Cardiovascular Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: A three-way randomized controlled crossover study will investigate the effects of fermented plant-based foods, non-fermented plant-based foods and the habitual diet on cardiometabolic risk factors. Each intervention will be ongoing for six weeks with six weeks washout in-between. During the fermented/non-fermented plant-based foods intervention, participants will add several corresponding food products to their habitual diet. The study has been dimensioned based on the estimated effect on hsCRP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fermented plant-based foods (Experimental)
  Interventions: Dietary Supplement: Fermented plant-based foods
- Non-fermented plant-based foods (Active Comparator)
  Interventions: Dietary Supplement: Non-fermented plant-based foods
- Habitual diet (Other)
  Interventions: Other: Habitual diet

INTERVENTIONS:
Dietary Supplement: Fermented plant-based foods — Participants will daily consume five different types of fermented plant-based foods, in addition to their habitual diet.
  Arms: Fermented plant-based foods
Dietary Supplement: Non-fermented plant-based foods — Participants will daily consume five different types of non-fermented plant-based foods, in addition to their habitual diet.
  Arms: Non-fermented plant-based foods
Other: Habitual diet — Participants will follow their habitual diet.
  Arms: Habitual diet

SUMMARY:
The primary objective of this study is to evaluate the metabolic effects of a high-fiber portfolio diet based on fermented plant-based foods compared to a corresponding non-fermented plant-based diet and a control diet (habitual diet). This will be assessed across gut microbiome profiles (high/low Prevotella), focusing on cardiometabolic risk factors, particularly inflammation.

A total of 100 men and women who meet all inclusion criteria and none of the exclusion criteria will be invited to participate. The study will employ a three-way randomized, controlled cross-over design, featuring six-week interventions separated by six-week washout periods. Participants will attend the clinic on 15 occasions, including screening visits.

ELIGIBILITY:
Inclusion Criteria:

* Sign of metabolic syndrome

Waist circumference > 102 cm/88 cm M/W and at least one of the following:

* High density lipoprotein (HDL) ≤1.0 mmol/L men / HDL ≤1.3 mmol/L
* Triglycerides ≥ 1,7 mmol/L
* Blood pressure ≥130/85 mmHg
* Fasting glucose ≥5.6 mmol/L

Other inclusion criteria:

* Signed informed consent
* Willingness to consume the intervention foods
* Body mass index 25-35 kg/m2
* Hemoglobin 120-160 g/L
* Serum thyroid-stimulating hormone (S-TSH) <4 mIU/L
* Serum C-reactive protein (S-CRP) <5 mg/L
* Access to a -18⁰ C freezer
* Any medication stable for the last 14 days.

Exclusion Criteria:

* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study.
* Following any weight reduction program or having followed one during the last 6 months
* Food allergies or intolerances
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption, colostomy, bowel resection, gastric bypass surgery, Helicobacter infection, Peptic ulcer disease, untreated celiac disease, etc.)
* Previous major gastrointestinal surgery
* Pregnant or lactating or wish to become pregnant during the period of the study.
* Unable to understand written and spoken Swedish
* Lack of suitability for participation in the trial, for any reason, as judged by the medical doctor or PI.
* Pharmacological medication with drugs known to affect the microbiota, e.g., antibiotics, within 6 months prior to baseline.
* Intake of any probiotic pills or foods enriched in probiotics within 6 months prior to baseline.
* Type I diabetes
* Small bowel bacterial overgrowth
* Diarrheal disease
* Receiving pharmacological treatment for type II diabetes (treatments based on lifestyle interventions are acceptable, as long as it is compatible with the study protocol)
* Using nicotine products on a daily basis (including chewing gum, patches, snus etc.)
* History of heart failure or heart attack (TIA) within 1 year prior to screening
* Thyroid disorder
* Planned surgery within the next eight months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
C-reactive protein | 6 weeks
  Investigate if c-reactive protein differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.

SECONDARY OUTCOMES:
Glucose | 6 weeks
  Investigate if glucose differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Insulin | 6 weeks
  Investigate if insulin differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Liver parameters | 6 weeks
  Investigate if liver parameters differ between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Glycaemic variability | 2 weeks
  Investigate if glycaemic variability differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Mixed meal tolerance test | 1-day
  Investigate if a mixed meal tolerance test causes different metabolic responses for the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet
Gut microbiome | 6 weeks
  Investigate if the fecal microbiome differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Blood pressure | 6 weeks
  Investigate if blood pressure differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Blood lipid profile | 6 weeks
  Description: Investigate if c-reactive protein differs between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.

OTHER OUTCOMES:
The metabolome | 6 weeks
  Investigate if the fecal, blood and urine metabolome differ between the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.
Gut microbiome profiles | 6 weeks
  Investigate if the response to the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet depends on the gut microbiome profile high/low Prevotella.
Transit time | 5-days
  Investigate if transit time, measured by intake of sweet corn, differs for the interventions fermented plant-based foods, non-fermented plant-based foods and the habitual diet.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard Landberg, PhD, Principal Investigator — Chalmers Univeristy of Technology
Locations (1):
- Sahlgrenska University Hospital, Wallenberg Lab, Gothenburg, Ästra Götaland, Sweden